CLINICAL TRIAL: NCT02806050
Title: Early Identification of Patients Who Benefit From Palbociclib in Addition to Letrozole
Brief Title: Palbociclib and FES PET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, C.P. Schroder, Principal investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201600066
Record Dates: First submitted 2016-05-17; First posted 2016-06-20 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: FES PET; Palbociclib
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib and FES PET (Experimental): To evaluate whether low uptake on FES-PET at baseline is related to non-response to letrozole plus palbociclib treatment.
  Interventions: Drug: Palbociclib; Device: FES PET; Drug: Letrozole

INTERVENTIONS:
Drug: Palbociclib — all patients will be treated with palbociclib, on a 3 weeks on, 1 week off cycle until progression
Device: FES PET — all patients will have a FES PET at baseline
Drug: Letrozole — all patients will be treated with Letrozole daily until progression

SUMMARY:
The purpose is to evaluate whether non invasive in vivo imaging of the estrogen receptor (ER) presence in metastatic breast cancer patient by means of 18F-fluoro-estradiol (FES) positron emission tomography (PET) can be used to predict treatment response to palbociclib plus letrozole. As ER expression predicts response to palbociclib in metastatic breast cancer patients the investigators hypothesize that lesions with low uptake on FES-PET will not respond to the combination of letrozole plus palbociclib.

DETAILED DESCRIPTION:
To evaluate in a feasibility study whether low uptake on FES-PET at baseline is related to non response to letrozole plus palbociclib treatment. The investigators will perform this feasibility study in 15 patients with metastatic breast cancer, eligible for letrozole and palbociclib therapy.

All patients will be treated with letrozole 2.5mg daily continuously throughout a 28-day cycle. This is combined with palbociclib 125 mg daily for 21 consecutive days followed by 7 days off treatment. At baseline all patients will have a FES PET scan. Currently the combination with palbociclib and letrozole has been approved by the FDA as initial endocrine-based therapy for postmenopausal women with ER positive HER2 negative advanced breast cancer. This is based on improved progression free survival with 10 months compared to endocrine therapy alone in both first and second line hormonal treatment for ER-positive metastatic breast cancer. In Europe, approval is expected late 2016. Therefore, in this study, all patients will receive a (presumably effective) treatment combination, that patients do not have standard access to in the Netherlands yet. In addition to the standard control visits to the clinic, two extra visits will be performed as part of the study: for screening and for the FES-PET scan. In the future, this study may potentially contribute to improved selection of patients for this combination treatment. This is of relevance in view of optimal treatment for individual patients, avoiding unnecessary toxicity and financial burden.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

1. Patients with ER positive (i.e. >1% staining), HER2 negative metastatic breast cancer (preferably assessment on fresh metastasis biopsy, alternatively archival metastasis biopsy)
2. Post-menopausal status defined as:

   * Age ≥60 years
   * Previous bilateral oophorectomy
   * Age <60 years and amenorrhea for >12 months in the absence of interfering hormonal therapies (such as LH-RH agonists and ER-antagonists
   * Age <60 years using ER antagonists should have amenorrhea for >12 months and FSH >24U/L and LH>14U/L
3. Adequate bone marrow and organ function defined as follows:

   * Absolute neutrophil count > 1.5 x 109/L
   * Platelet count >100 x 109/L
   * White blood cell count >3 x 109/L
   * AST and ALT <3.0 x upper limit of normal (ULN) or <5 xULN in case of known liver metastases.
   * Alkaline phosphatase <2.5 x ULN
   * Total serum bilirubin < ULN or total bilirubin <3.0 x ULN with direct bilirubin within normal range in patients with Gilbert's Syndrome
   * Creatinine clearance >50mL/min
   * Lipase/amylase <1/5 x ULN
   * Prothrombin time, partial thromboplastin time and INR <1.5 x ULN
4. ECOG performance 0-2
5. Signed written informed consent
6. Able to comply with the protocol
7. Age ≥18 years

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Life expectancy < 3 months
2. Evidence of central nervous system metastases
3. Presence of life-threatening visceral metastases
4. Prior use of CDK4/6 inhibitor
5. Use of estrogen receptor ligands including estrogens, fulvestrant or tamoxifen <6 weeks before study entry.
6. Use of other anticancer therapy < 2 weeks prior to start with palbociclib
7. Concurrent malignancy
8. Active cardiac disease or a history of cardiac dysfunction
9. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to the start of treatment that are known strong inducers or inhibitors of CYP3A4/5, known risk to prolong the QT interval or induce Torsades de Pointes, or narrow therapeutic window and are predominantly metabolized through CYP3A4/5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
The relation between low uptake on FES-PET to response per lesion | 8 weeks after start of treatment

SECONDARY OUTCOMES:
quantitative FES-uptake and correlation with progression free survival | 6 months
analysis of circulating tumor DNA and correlation with FES-PET results and progression free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: C. P. Schröder, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boers J, Venema CM, de Vries EFJ, Glaudemans AWJM, Kwee TC, Schuuring E, Martens JWM, Elias SG, Hospers GAP, Schroder CP. Molecular imaging to identify patients with metastatic breast cancer who benefit from endocrine treatment combined with cyclin-dependent kinase inhibition. Eur J Cancer. 2020 Feb;126:11-20. doi: 10.1016/j.ejca.2019.10.024. Epub 2019 Dec 28. PMID 31891878